CLINICAL TRIAL: NCT04356430
Title: Medical Ethics Committee of Nanjing Drum Tower Hospital Affiliated to Medical School of Nanjing University
Brief Title: Neoadjuvant Therapy of Abiraterone Plus ADT for High Risk Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Director of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-101
Record Dates: First submitted 2020-04-12; First posted 2020-04-22 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; Goserelin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADT with Abiraterone and prednisone (Experimental): All subjects in this arm will receive luteinizing hormone releasing hormone analogue (LHRHa) plus abiraterone acetate and prednisone, as per standard of care. Goserelin 10.8 mg will be used once per 12 weeks. Abiraterone acetate will be administered orally as 1000 mg once daily along with 5 mg of oral prednisone once per day. Subjects will continue to take abiraterone acetate and prednisone for 24 weeks before robotic assisted radical prostatectomy
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone; Drug: Goserelin 10.8 mg
- ADT alone (Experimental): All subjects in this arm will receive LHRHa alone for 24 weeks before receiving robotic assisted radical prostatectomy. Goserelin 10.8 mg will be administered once per 12 weeks.
  Interventions: Drug: Goserelin 10.8 mg

INTERVENTIONS:
Drug: Abiraterone Acetate — 1000 mg orally daily for 24 weeks before robotic assisted radical prostatectomy
  Arms: ADT with Abiraterone and prednisone
Drug: Prednisone — 5 mg oral low dose prednisone, once daily
  Arms: ADT with Abiraterone and prednisone
Drug: Goserelin 10.8 mg — 10.8 mg goserelin hypodermic once per 12 weeks

SUMMARY:
High risk prostate cancer (PCa) had worse outcomes on radical treatment results, short-time oncological results, even cancer-specific survival, than those low or mediate risk PCa. Neoadjuvant treatment before radical prostatectomy had been proven to get some benefits on peri-operation results, especially on reduction of tumor volume and minimization of biochemical recurrence. This study will evaluate the efficacy and safety of androgen deprivation therapy (ADT) with abiraterone in neoadjuvant therapy for surgically resectable high-risk or very high-risk PCa.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 and ≤75 years of age.
* All patients must have a histologically or cytologically diagnosis of prostate cancer and must be eligible for radical prostatectomy.
* All patients must undergo thorough tumor staging and meet one of the following criteria: 1. multi-parameter MRI or PSMA PET / CT shows clinical staging of primary tumor ≥ T3, 2. Gleason score of primary tumor ≥ 8, 3. prostate specific antigen (PSA) ≥20 ng/ml.
* Eastern Cooperative Oncology Group (ECOG) physical condition score ≤ 1
* Patients must have adequate hematologic function, within 28 days prior to registration as evidenced by: white blood cell (WBC) ≥ 4.0 × 109 / L, platelets≥ 100 × 109 / L, hemoglobin ≥ 9 g / dL, and international normalized ratio (INR) < 1.5.
* Patients must have adequate hepatic function, within 28 days prior to registration, as evidenced by: total bilirubin (TBIL)≤1.5 x upper limit of normal (ULN),and SGOT (AST) and SGPT (ALT) ≤ 2.5 x ULN.
* Patients must have adequate renal function, within 28 days prior to registration, as evidenced by serum creatinine ≤2×ULN
* Patients must participate voluntarily and sign an informed consent form (ICF), indicating that they understand the purpose and required procedures of the study, and are willing to participate in. Patients must be willing to obey the prohibitions and restrictions specified in the research protocol.

Exclusion Criteria:

* Patients with prostate having neuroendocrine, small cell, or sarcoma-like features are not eligible.
* Patients with low-risk and medium-risk, localized prostate cancer (the following conditions are met at the same time) are not eligible: multi-parameter MRI or PSMA PET / CT shows clinical staging of primary tumor < T3, Gleason score of primary tumor < 8, and prostate specific antigen (PSA) <20 ng/ml.
* Patients with clinical or radiological evidence of regional or extra-regional lymph node metastases or bone metastases or visceral metastases are not eligible.
* Patients with clinical or radiological evidence of regional or extra-regional lymph node metastases or bone metastases or visceral metastases are not eligible.
* Patients who have previously received androgen deprivation therapy (medical or surgical) or focal treatment of prostate cancer or prostate cancer radiotherapy or prostate cancer chemotherapy are not eligible.
* Patients with severe or uncontrolled concurrent infections are not eligible.
* Patients must not have New York Heart Association Class III or IV congestive heart failure at the time of screening. Patients must not have any thromboembolic event, unstable angina pectoris, myocardial infarction within 6 months prior to registration.
* Patients must not have uncontrolled severe hypertension, persistent uncontrolled diabetes, oxygen-dependent lung disease, chronic liver disease, or HIV infection.
* Patients must not have had other malignancies other than prostate cancer in the past 5 years, but cured basal cell or squamous cell skin cancers can be enrolled.

Patients with mental illness, mental disability or inability to give informed consent are not eligible.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate | up to 8 months
  The proportion of subjects with no morphologically recognizable cancer cell in tumor specimens after radical prostatectomy
Proportion of Subjects With Minimal Residual Disease | up to 8 months
  The proportion of subjects that have residual tumors with maximum diameter of 5 mm or less after radical prostatectomy

SECONDARY OUTCOMES:
Rate of Stage Degradation | up to 8 months
  Clinical or pathological stage degradation after neoadjuvant therapy
Rate of Positive Surgical Margins | up to 8 months
  The proportion of subjects with positive surgical margins after radical prostatectomy
Rate of Complete Serum Remission | up to 6 months
  The proportion of subjects whose PSA is less than or equal to 0.2 ng/ml after 6 months of treatment
Proportion of subjects without PSA progression | 24 months
  The proportion of subjects whose PSA has never gone below 1 ng/ml or who receive any radiotherapy or systemic treatment after radical prostatectomy
Imaging Response Rate | up to 8 months
  The proportion of subjects whose primary tumor is in complete remission on imaging or residual tumor's maximum diameter is less than 0.5cm
Recovery time of urinary continence (day) | 12 month
  The recovery time of urinary continence (day) after radical prostatectomy, defined as 0 pad/day.
biochemical recurrence-free survival (bRFS) | 3 years
  biochemical recurrence-free survival (bRFS) defined as time to PSA ≥ 0.2 ng/ml after radical prostatectomy.
metastasis-free survival (MFS) | 5 years
  time from date of randomization to date of evidence of systemic disease on bone scan or cross-sectional imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, MD, Principal Investigator — Nanjing Drum Tower Hospital, affiliated to medical school of Nanjing University
Locations (1):
- Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhuang J, Wang Y, Zhang S, Fu Y, Huang H, Lyu X, Zhang S, Marra G, Xu L, Qiu X, Guo H. Androgen deprivation therapy plus abiraterone or docetaxel as neoadjuvant therapy for very-high-risk prostate cancer: a pooled analysis of two phase II trials. Front Pharmacol. 2023 Jun 26;14:1217303. doi: 10.3389/fphar.2023.1217303. eCollection 2023. PMID 37435500